CLINICAL TRIAL: NCT06226350
Title: An Open, Single-arm, Multicenter Phase II Trial of Efficacy and Safety of F520 Monotherapy in the Treatment of Advanced, Persistent, Recurrent, or Metastatic Cervical Cancer
Brief Title: A Phase Ⅱ Study of F520 in Patients With Cervical Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTP-F520-005
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- F520 monotherapy (Experimental)
  Interventions: Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection

INTERVENTIONS:
Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection — F520,IV, 3mg/kg every 3 weeks, for up to 2 years until disease progression, intolerable toxic reactions, or termination of treatment for other reasons.

SUMMARY:
This study was an open, single-arm, enriched, multicenter Phase II study.

DETAILED DESCRIPTION:
The trial was divided into screening period, treatment period and follow-up period. Participants entered the screening period after signing informed consent and met the inclusion criteria. Subjects who did not meet the exclusion criteria were treated with F520 monotherapy, intravenously, at 3mg/kg every 3 weeks until disease progression or intolerable toxicity or withdrawal for other reasons, for a maximum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years and above;
2. Cervical squamous cell carcinoma, adenosquamous cell carcinoma or adenocarcinoma confirmed by histopathology;
3. Patients with advanced (stage IVb) cervical cancer that is inoperable and/or radiotherapy-resistant, or patients with persistent, recurrent or metastatic cervical cancer that progresses after first-line or above chemotherapy;
4. According to RECIST1.1 criteria, subjects must have at least one measurable target lesion examined by enhanced CT and/or enhanced MRI (non-lymph node diameter ≥10mm, or lymph node lesion diameter ≥15mm);
5. Expected survival ≥3 months;
6. Those with 0-2 scores on the American Eastern Oncology Collaboration Group (ECOG) scale;
7. Those who agree to provide archived tumor tissue samples or fresh tissue samples;
8. The function of vital organs meets the following requirements (drugs with blood components and cell growth factors are not allowed to be used within 14 days before the first administration) :

Blood routine: Absolute neutrophil count ≥1.5×109/L; Platelet ≥75×109/L; Hemoglobin ≥90g/L; Liver function: TBIL≤1.5×ULN, ALT and AST≤2.5×ULN; If liver metastasis was present, TBIL≤3×ULN, ALT and AST≤5×ULN; Renal function: serum creatinine (Cr) ≤1.5×ULN; Thyroid stimulating hormone (TSH) in the normal range; If TSH is abnormal, free triiodothyronine (FT3) and free thyroxine (FT4) must be normal or abnormal without clinical significance.

International Normalized ratio (INR) ≤1.5×ULN and activated partial thromboplastin time (APTT) ≤1.5×ULN.

Exclusion Criteria:

1. Patients with specific pre-existing conditions such as active autoimmune disease, type 1 diabetes, hypothyroidism requiring hormone replacement, and severe mental illness;
2. a history of other malignancies within the last 3 years, except locally curable cancers (limited to basal cell or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the breast);
3. Patients with central nervous system metastasis with clinical symptoms;
4. Previously treated with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibodies or any other antibody or drug targeting T-cell co-stimulation or immune checkpoint pathways;
5. Immunosuppressive, systemic or local hormone therapy within 14 days prior to initial administration for immunosuppressive purposes (daily dose equivalent to prednisone > 10mg of systemic corticosteroid);
6. Active infection requiring systemic treatment or unexplained fever during screening or prior to initial dosing > 38.5℃ (according to the investigators' judgment, patients with fever caused by tumors could be included in the group);
7. Patients receiving systemic tumor therapy with radiotherapy, chemotherapy, hormone therapy, surgery, targeted therapy or antibody drugs within 4 weeks before the first dose; Those who had been treated with monoclonal antibody coupled radionuclides or cytotoxins within 10 weeks prior to initial administration; The toxicity of previous anti-tumor therapy did not return to ≤ grade 1 (except hair loss);
8. Those who have had previous organ transplantation or received autologous stem cell transplantation within 3 months before the first administration;
9. infected with active tuberculosis;
10. suffering from interstitial lung disease (except for interstitial lung disease caused by radiotherapy and chemotherapy and currently asymptomatic);
11. Active hepatitis;
12. HIV antibody positive;
13. have been treated with any other investigational drug/device within 4 weeks prior to initial dosing;
14. Have uncontrolled or severe cardiovascular disease, such as New York Heart Association (NYHA) Class II or above congestive heart failure, unstable angina, myocardial infarction and other cardiovascular disease within 6 months before the first dose; Difficult to control hypertension (systolic blood pressure ≥180mmHg and/or diastolic blood pressure ≥100mmHg);
15. Those who have a history of drug abuse or alcoholism within 6 months before the first dose;
16. Known patients with previous macromolecular protein preparations, or known anti-PD-1 /PD-L1 antibodies;
17. Those who received live attenuated vaccine within 4 weeks prior to the first dose (except inactivated influenza vaccines such as injectable seasonal influenza vaccine);
18. Pregnant or lactating women, women who planned to become pregnant during the study period and within 6 months after the last dose, and who did not wish to use a medically approved effective contraceptive method (such as an IUD or condom) during the trial period;
19. Those who were judged not suitable for inclusion by the researchers.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Objective tumor response rate (ORR) assessed by RECIST1.1 | approximately 2 years
  CR+PR

CONTACTS AND LOCATIONS:
Overall Officials: QI ZHOU, MD, Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Shandong New Time Pharmaceutical Co., LTD, Shandong, China